CLINICAL TRIAL: NCT01211366
Title: Post-operative Infusion of Intra-operative Cell Salvage Reduces Allogeneic Blood Product Transfusions and Volume Resuscitation in Pediatric Cardiac Surgery and Improves Clinical Outcomes
Brief Title: Use of Cell Salvage Post-operatively in Infants to Decrease Use of Allogeneic Blood Product Transfusions
Acronym: cell salvage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, jill cholette, Assistant Professor of Pediatrics, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 32600
Record Dates: First submitted 2010-09-28; First posted 2010-09-29 (Estimated); Last update posted 2012-02-13 (Estimated); Status verified 2012-02

CONDITIONS: Transfusion
Keywords: cell saver; allogeneic RBCs; washed cells; PRBC transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional Transfusion (Active Comparator): Infants will receive PRBCs, crystalloid, and colloid for hemodynamic instability per the usual routine at the discretion of the attending intensive care physician
  Interventions: Other: Conventional volume infusion
- Cell Saver (Experimental): Infants will receive washed cell-saver RBCs for hemodynamic instability in the first 24 hours post-operative period as long as Hgb is < 13 gm/dL and cell-saver is available.
  Interventions: Other: Cell Saver RBCs

INTERVENTIONS:
Other: Cell Saver RBCs — Use of cell saver RBCs to decrease the infusion of allogeneic PRBCs, crystalloid, and colloid in post-operative infants following CPB as needed for hemodynamic instability
  Arms: Cell Saver
Other: Conventional volume infusion — Infusion of allogeneic PRBCs, crystalloid, and colloid as needed for hemodynamic instability
  Arms: Conventional Transfusion

SUMMARY:
Transfusion of washed intra-operative cell salvage post-operatively in the PCICU can be performed safely without increased risk of bleeding or release of inflammatory mediators. This will reduce the need for allogeneic blood products as well as crystalloid and colloid infusions and thus decrease the length of ventilation and intensive care duration for these infants.

ELIGIBILITY:
Inclusion Criteria:

* 1. Weight < or = 20Kg;
* 2. Cardiac surgery with CPB at URMC;
* 3. informed consent

Exclusion Criteria:

* 1. weight > 21 Kg;
* inability to obtain consent;
* non-English speaking

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2010-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Comparison of volume of allogeneic blood products and crystalloid/colloid infusions between groups | 2 years
  To compare the volume of allogeneic blood products and crystalloid/colloid infusions between patients randomized to receive washed intra-operative cell salvage vs our current standard for volume replacement for the first 24 hours post-op

SECONDARY OUTCOMES:
comparison of bleeding, use of coagulant products, and inflammatory markers between groups | 2 years
  To compare measures of bleeding (MT drainage, Hgb, platelet counts) , the use of coagulant products (FFP, platelets, cryoprecipitate) and inflammatory/immunomodulatory markers [C-reactive protein (CRP) and IL-6/IL-10 ratio]between patients randomized to receive washed intra-operative cell salvage vs our current standard of care for volume replacement.
comparison of clinical outcomes between groups | 2 years
  To compare clinical outcome measures (ventilator days, PCICU duration, thrombosis, bacterial infections and mortality) between patients randomized to receive washed intra-operative cell salvage vs our current standard of care for volume replacement.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States